CLINICAL TRIAL: NCT03474354
Title: Correlation of Necrosis With DC Bead LUMI (TM) Distribution
Brief Title: DC Bead LUMI (TM) Loaded With Doxorubicin for Intermediate Hepatocellular Carcinoma (HCC)
Status: Completed | Type: Observational
Sponsor: Malagari Katerina (Other)
Responsible Party: Sponsor-Investigator, Malagari Katerina, ASSOCIATE PROFESSOR, University of Athens
Organization: University of Athens (Other)
Other Study IDs: IIS_Malagari Athens_BTG
Record Dates: First submitted 2018-02-13; First posted 2018-03-22 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Hepatocellular Cancer; Chemoembolization
Keywords: chemoembolization; drug eluting beads
MeSH Terms: conditions — Liver Neoplasms | interventions — Chemoembolization, Therapeutic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: chemoembolization — correlation of necrosis with the deposition of beads

SUMMARY:
The primary purpose of the study is to evaluate the distribution of radiopaque microspheres loaded with doxorubicin in the treatment of unresectable HCC. Prospective, single arm, open label, single centre, pilot study. All patients will undergo clinical follow-up. Twenty patients will be enrolled.

DETAILED DESCRIPTION:
The primary purpose of the study is to evaluate the distribution of radiopaque microspheres loaded with doxorubicin in the treatment of unresectable HCC. Prospective, single arm, open label, single centre, pilot study. All patients will undergo clinical follow-up. Twenty patients will be enrolled. Primary endpoint : Local response (evaluated with CT and MRI at 4 to 6 weeks post each procedure and at 6 months according to mRECIST) in patients with intermediate-stage HCC following chemoembolisation with radiopaque bead. Secondary endpoints include: 1) Better definition of end point of embolization for drug eluting beads : Ability to achieve near-stasis during chemoembolisation procedure in the tumour feeding vessels using intra-procedural imaging feedback from the radiopaque bead (early visualization of non target embolization 2) Total dose needed for tumor devascularization 3)Distribution of radiopaque beads and correlation with necrosis and adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old.
2. HCC diagnosed according to updated American Association for the Study of Liver Diseases (AASLD) criteria.
3. Barcelona Criteria Liver Cancer (BCLC) stage B patients or BCLC stage A patients not candidates for curative treatment (resection, transplantation, ablation) or who have failed/recurred after resection/ablation).
4. Tumour burden (located in one or two lobes) that can be sufficiently and selectively embolised with required dose or radiopaque bead loaded with doxorubicin.
5. Performance status: Eastern Cooperative Oncology Group (ECOG) status 0/1.
6. Normal liver or compensated cirrhosis with preserved liver function (Child-Pugh A score and Child/Pugh B≤ 7 points ) without ascites.
7. Total bilirubin ≤2.0 mg/dl.
8. Adequate renal function (serum creatinine < 1.5 X ULN).
9. Patient has provided written informed consent.

Exclusion Criteria:

1. Patient previously treated with any intra-arterial therapy for HCC.
2. Eligible for curative treatment (resection/RadioFrequency Ablation-RFA, transplantation therapies).
3. Advanced liver disease: Child-Pugh's C class or active gastrointestinal bleeding, encephalopathy. Bilirubin levels >2.0 mg/dl.
4. Advanced tumoural disease: BCLC class C (vascular invasion -even segmental, extra-hepatic spread or cancer-related symptoms=ECOG of 1-2) or D class (WHO performance status 3 or 4, Okuda III stage).
5. Patient with another primary tumour.
6. Patient with refractory ascites or on diuretic treatment; minor ascites retention detected at imaging and not requiring diuretics to be solved is not a contraindication.
7. Patient with history of biliary tree disease or biliary dilatation.
8. Portal vein thrombosis, porto-systemic shunt, hepatofugal blood flow or absent portal blood flow in the liver area to be treated.
9. Contraindication to multiphasic CT and MRI (e.g. allergy to contrast media).
10. Any other contraindication for embolisation or local doxorubicin treatment.
11. Patients currently receive treatment with any investigational drug/device/intervention or have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) before study treatment.
12. In the Investigator's opinion patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
13. Pregnant or breast-feeding women.

Ages: 18 Years to 88 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate stage hepatocellular carcinoma (BCLC B)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
CORRELATION OF LUMI DISTRIBUTION WITH NECROSIS | 12 months
  Local response following chemoembolisation

SECONDARY OUTCOMES:
Definition of end point of embolization for drug eluting beads | 12 months
  optimization of embolization
Total dose needed for tumor devascularization | 12 months
  dose required for tumor devascularization
Distribution of radiopaque beads and correlation with necrosis | 12 months
  correlation between imaging and tumor necrosis

CONTACTS AND LOCATIONS:
Overall Officials: KATERINA MALAGARI, Principal Investigator — Evgenidion Hospital Athens, Greece
Locations (1):
- Evgenidion Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Yes
CT and MRI images will be stored anonymously by giving each patient a code number
Supporting Information: CSR
Time Frame: starting February 2018 and ending February 2019
Access Criteria: the principal investigator and collaborator will record and analyse data from the CT and MRI of the patients. The names of the patients will not be in the examinations and identity will be given by enrollment number